CLINICAL TRIAL: NCT06194955
Title: The Effect of Glucose-dependent Insulinotropic Polypeptide (GIP), Glucagon-like Peptide-1 (GLP-1) and Glucagon-like Peptide-2 (GLP-2) in Individuals With Genetically Altered Receptor Function
Brief Title: The Effect of GIP, GLP-1 and GLP-2 in Individuals With Genetically Altered Receptor Function
Acronym: H-21044858
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Gentofte Hospital, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-21044858
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Incretin Effect
Keywords: Gut hormones; single nucleotide variants (SNVs); GIP; GLP-1; GLP-2
MeSH Terms: interventions — gastric inhibitory polypeptide (1-42); Glucagon-Like Peptide 1

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized, crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GIPR variant carriers (Active Comparator): Inidividuals with GIPR variants: Determination of the incretin effect, and the insulinotropic actions of GIP and GLP-1 infusions during hyperglycemic clamp.
  Interventions: Drug: GIP(1-42); Drug: GLP-1; Other: Placebo
- GIPR variant carrier controls (Placebo Comparator): Healthy matched individuals: Determination of incretin effect, and the insulinotropic actions of GIP and GLP-1 infusions during hyperglycemic clamp.
  Interventions: Drug: GIP(1-42); Drug: GLP-1; Other: Placebo
- GLP-1R variant carrier (Active Comparator): Individuals with GLP-1R variants: Determination of incretin effect, and the insulinotropic actions of GIP and GLP-1 infusions during hyperglycemic clamp
  Interventions: Drug: GIP(1-42); Drug: GLP-1; Other: Placebo
- GLP-1R variant carrier controls (Placebo Comparator): Healthy matched individuals: Determination of incretin effect, and the insulinotropic actions of to GIP and GLP-1 infusions during hyperglycemic clamp.
  Interventions: Drug: GIP(1-42); Drug: GLP-1; Other: Placebo
- GLP-2R variant carrier (Active Comparator): Individuals with GLP-2R variants: Determination of bone resorption marker levels (CTX) and response to GLP-2 infusions during fasting blood glucose levels
  Interventions: Drug: GLP-2; Other: Placebo
- GLP-2R variant carrier control (Placebo Comparator): Healthy matched individuals: Determination of bone resorption marker levels (CTX) and response to GLP-2 infusions during fasting blood glucose levels
  Interventions: Drug: GLP-2; Other: Placebo

INTERVENTIONS:
Drug: GIP(1-42) — Infusion
  Arms: GIPR variant carrier controls; GIPR variant carriers; GLP-1R variant carrier; GLP-1R variant carrier controls
Drug: GLP-1 — Infusion
  Arms: GIPR variant carrier controls; GIPR variant carriers; GLP-1R variant carrier; GLP-1R variant carrier controls
Drug: GLP-2 — Infusion
  Arms: GLP-2R variant carrier; GLP-2R variant carrier control
Other: Placebo — Saline

SUMMARY:
This project will characterize the physiological effect of the hormones, GIP-, GLP-1- and GLP-2 infusions in a group of individuals that are carriers of GIP-, GLP-1- and GLP-2 receptor gene variants, respectively.

DETAILED DESCRIPTION:
Participants with mutations in their GLP-1- and GIP receptor will attend five randomized experimental days, A1, A2, B, C and D. On day A1 an oral glucose tolerance test (OGTT) will be performed, and on day A2, an intravenous isoglycaemic glucose infusion (IIGI) will be performed. On experimental day B and C, the study participants will receive GLP-1 and GIP hormones, respectively, under stable glucose infusions and on experimental day D, they will receive infusion of salt water (placebo) under stable glucose infusion.

Participants with mutations in their GLP-2 receptor will attend three randomized experimental days, E, F and G. A mixed meal test (MMT) will be performed on day E, an infusion with GLP-2 during fasting blood glucose levels will be performed on day F, and infusion with salt water (placebo) during fasting blood glucose levels will be performed on day G.

Additionally, a DXA scan and arginine test will be performed on all study participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-35 kg/m2

Exclusion Criteria:

* Treatment with medication or supplements that can not be discontinued for 12 hours
* >10 objects of alcohol weekly or abuse of narcotics
* Liver disease (defined as ALAT and/or ASAT ≥ 2 x normal levels)
* Decreased kidney function (creatine levels over reference interval)
* Uncontrollable increased blood pressure (> 140/90 mmHg)
* Low blood percentage (hemoglobin < 8.3 mmol/l)
* Special diet or planned weight change during trial period
* Other conditions that could be expected to affect the primary or secondary outcomes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
For GIP- and GLP-1 receptor variants: Insulinotropic effect (C-peptide) | 240 minutes
  Blood sample
For GLP-2 receptor variants: CTX (bone resorption marker) | 120 minutes
  Blood sample

SECONDARY OUTCOMES:
GIP levels | 240 minutes
  Blood sample
GLP-1 levels | 240 minutes
  Blood sample
GLP-2 levels | 240 minutes
  Blood sample
CTX (bone resorption marker) | 240 minutes
  Blood sample
P1NP (bone formation marker) | 240 minutes
  Blood Sample
Heart rate | 240 minutes
  Beats/minute
Insulin | 240 minutes
  Blood sample
Glucagon | 240 minutes
  Blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes